CLINICAL TRIAL: NCT03540823
Title: Immunogenicity and Safety of Influenza A/H3N2 Vaccine in Patients With Rheumatologic Diseases
Brief Title: Evaluation of Influenza A/H3N2 Vaccine in Patients With Rheumatologic Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H3N2VaccineReumatoHC
Record Dates: First submitted 2018-05-14; First posted 2018-05-30 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-04

CONDITIONS: Systemic Lupus; Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with rheumatic diseases (Experimental): Patients with diagnosis of adult and juvenile systemic lupus erythematosus (SLE and JSLE) and Sjogren syndrome (SSp)
  Interventions: Biological: Inactivated and fragmented influenza vaccine (A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus)
- Healthy controls (Other): Healthy children and adults
  Interventions: Biological: Inactivated and fragmented influenza vaccine (A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus)

INTERVENTIONS:
Biological: Inactivated and fragmented influenza vaccine (A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus) — Single dose of Inactivated and fragmented influenza vaccine (A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus)

SUMMARY:
Studies in the literature have shown reduced effectiveness of influenza A (H3N2) virus vaccine (20-40%) when compared to A (H1N1) and influenza B. This reduction in efficacy may partly result of the need to propagate A (H3N2) virus into egg components for the preparation of the vaccine. Other factors that may also contribute to the reduction of efficacy against A (H3N2) viruses include the high level of genetic diversity and the rate of rapid evolution of this particular virus subtype and the modification of the immune response to the vaccine secondary of prior infection or vaccination.

Vaccine efficacy studies are required to verify the immunogenicity of the H3N2 influenza vaccine in immunosuppressed patients with rheumatologic disease. In addition, it is relevant to evaluate the safety of the vaccine in this population as well as the possibility of reactivation of the rheumatologic disease itself. The objectives of this study are to evaluate the immunogenicity of the H3N2 component of the inactivated and fragmented influenza vaccine in patients with two systemic autoimmune rheumatic diseases (Systemic Lupus Erythematosus - Adult and Juvenile, Primary Sjögren's Syndrome).

DETAILED DESCRIPTION:
Studies in the literature have shown reduced effectiveness of influenza A (H3N2) virus vaccine (20-40%) when compared to A (H1N1) and influenza B. This reduction in efficacy may partly result of the need to propagate A (H3N2) virus into egg components for the preparation of the vaccine. Other factors that may also contribute to the reduction of efficacy against A (H3N2) viruses include the high level of genetic diversity and the rate of rapid evolution of this particular virus subtype and the modification of the immune response to the vaccine secondary of prior infection or vaccination.

Vaccine efficacy studies are required to verify the immunogenicity of the H3N2 influenza vaccine in immunosuppressed patients with rheumatologic disease. In addition, it is relevant to evaluate the safety of the vaccine in this population as well as the possibility of reactivation of the rheumatologic disease itself. The objectives of this study are to:

1. Evaluate the immunogenicity of the H3N2 component of the inactivated and fragmented influenza vaccine (A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus] in patients with two systemic autoimmune rheumatic diseases (Systemic Lupus Erythematosus - Adult and Juvenile, Primary Sjögren's Syndrome).
2. Assess the safety of immunization with the inactivated influenza vaccine [A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus] in these patients with systemic autoimmune rheumatic diseases.
3. Evaluate the possible association between vaccinal immunogenicity with: demographic data, clinical and laboratorial activity of the disease, and treatment of patients with these rheumatic diseases.

Patients with diagnosis of adult and juvenile systemic lupus erythematosus (SLE and JSLE) (n=100) and Sjogren syndrome (SSp) (n=30) according to the classification criteria established for these diseases will be prospectively evaluated at the Hospital das Clínicas of the University of São Paulo (HC-FMUSP).

The control group will consist of 120 healthy individuals who will be recruited into the vaccination campaign paired for age and sex. The juvenile control group will be composed of 50 healthy children who will be recruited in the vaccination campaign paired for age and sex.

Patients and healthy controls will be vaccinated with one dose of the inactivated and fragmented influenza vaccine (A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus].

At study entry (D0) and after 30-45 days, blood sample will be collected from patients (SLE, SLE and SSp) and controls.

At entry (D0) and end of study (between D30-D45), patients will be assessed for clinical and laboratory disease activity through specific disease indexes of inflammatory activity: SLE: SLEDAI (lab: blood count, anti-dsDNA, complement, urine I and prot / creat ratio + 1 dry tube for H3N2 serology); SSp: EULAR Sjogren's syndrome disease activity index (Lab: PCR, anti-Ro / SS-A and anti-La / SS-B + 1 dry tube for H3N2 serology).

Patients and healthy controls are advised on possible side effects of the vaccine. In addition, patients and controls are instructed to note in a standardized diary symptoms during study period, such as pruritus, local pain, erythema, induration at the site of the vaccine, fever, chills, headache, myalgia, arthralgia and diarrhea. Signs of airway infections (cough, sputum, sore throat, nasal congestion or expectoration), fever (axillary temperature> 37.8 °C), need for hospitalizations, severity of infections, sick days, absenteeism at work, and treatment received for infections. Serious adverse events will be defined as those resulting in hospitalization or death. A contact telephone number for patients and controls is provided for guidance on moderate to severe adverse events.

Patients and controls are advised to contact the investigators in case of flu symptoms up to 6 months after vaccination to be evaluated clinically and with nasal swab collection for respiratory virus.

ELIGIBILITY:
Inclusion Criteria:

* Adult and juvenile systemic lupus erythematosus (SLE) and juvenile SLE patients according to the ACR classification criteria aged ≥ 18 years for adults and aged ≥ 9 and <18 years for the juvenile group
* Patients with primary Sjögren's Syndrome (SSp) (classification criteria of the European Study Group on Diagnostic Criteria for Sjögren's Syndrome) aged ≥ 18 years

Exclusion Criteria:

1. History of anaphylactic response to vaccine components or egg allergy
2. Moderate or severe acute febrile illness
3. Guillain-Barré syndrome, decompensated heart failure (class III or IV), demyelinating disease.
4. History of live virus vaccine up to 4 weeks before, virus vaccine inactivated up to 2 weeks prior, influenza vaccine up to 6 months prior to study.
5. History of having received blood products up to 6 months prior to the study.
6. Individuals who do not agree to participate in the study and / or whose parents do not agree to participate in the study.
7. Inpatients
8. Patients with severe conditions requiring hospitalization

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with seroprotection and seroconversion after Influenza vaccine | 30 days
  Immunogenicity (seroprotection and seroconversion) of the H3N2 component of the inactivated and fragmented influenza vaccine (A / Michigan / 45/2015 (H1N1) pdm09-like virus, A / Singapore / INFIMH-16-0019 / 2016 (H3N2) -like virus; B / Phuket / 3073/2013-like virus) will be evaluated by haemagglutination inhibition (HI) assay

SECONDARY OUTCOMES:
Number of participants with vaccine-related adverse events as assessed by CTCAE v4.0 | 30 days
  Patients and healthy controls are instructed to note all symptoms in a standardized diary during study period, such as pruritus, local pain, erythema, induration at the site of the vaccine, fever, chills, headache, myalgia, arthralgia and diarrhea. Signs of airway infections (cough, sputum, sore throat, nasal congestion or expectoration), fever (axillary temperature> 37.8 °C), need for hospitalizations, severity of infections, sick days, absenteeism at work, and treatment received for infections. Serious adverse events will be defined as those resulting in hospitalization or death. Number of participants with vaccine-related adverse events will be assessed by CTCAE v4.0 and the following reference: "Saad CG, Borba EF, Aikawa NE, et al. Immunogenicity and safety of the 2009 non-adjuvanted influenza A/H1N1 vaccine in a large cohort of autoimmune rheumatic diseases. Ann Rheum Dis. 2011;70:1068-73."

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Borba, MD, PhD, Principal Investigator — Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo São Paulo, Sao Paulo Brazil
Locations (1):
- Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva CA, Aikawa NE, Bonfa E. Vaccinations in juvenile chronic inflammatory diseases: an update. Nat Rev Rheumatol. 2013 Sep;9(9):532-43. doi: 10.1038/nrrheum.2013.95. Epub 2013 Jul 2. PMID 23820860
- [Background] Pasoto SG, Ribeiro AC, Bonfa E. Update on infections and vaccinations in systemic lupus erythematosus and Sjogren's syndrome. Curr Opin Rheumatol. 2014 Sep;26(5):528-37. doi: 10.1097/BOR.0000000000000084. PMID 25022358
- [Background] Kuruma KA, Borba EF, Lopes MH, de Carvalho JF, Bonfa E. Safety and efficacy of hepatitis B vaccine in systemic lupus erythematosus. Lupus. 2007;16(5):350-4. doi: 10.1177/0961203307078225. PMID 17576737
- [Background] Aikawa NE, Franca IL, Ribeiro AC, Sallum AM, Bonfa E, Silva CA. Short and long-term immunogenicity and safety following the 23-valent polysaccharide pneumococcal vaccine in juvenile idiopathic arthritis patients under conventional DMARDs with or without anti-TNF therapy. Vaccine. 2015 Jan 29;33(5):604-9. doi: 10.1016/j.vaccine.2014.12.030. Epub 2014 Dec 29. PMID 25554240
- [Background] Saad CG, Borba EF, Aikawa NE, Silva CA, Pereira RM, Calich AL, Moraes JC, Ribeiro AC, Viana VS, Pasoto SG, Carvalho JF, Franca IL, Guedes LK, Shinjo SK, Sampaio-Barros PD, Caleiro MT, Goncalves CR, Fuller R, Levy-Neto M, Timenetsky Mdo C, Precioso AR, Bonfa E. Immunogenicity and safety of the 2009 non-adjuvanted influenza A/H1N1 vaccine in a large cohort of autoimmune rheumatic diseases. Ann Rheum Dis. 2011 Jun;70(6):1068-73. doi: 10.1136/ard.2011.150250. PMID 21540203
- [Background] Aikawa NE, Campos LM, Silva CA, Carvalho JF, Saad CG, Trudes G, Duarte A, Miraglia JL, Timenetsky Mdo C, Viana VS, Franca IL, Bonfa E, Pereira RM. Glucocorticoid: major factor for reduced immunogenicity of 2009 influenza A (H1N1) vaccine in patients with juvenile autoimmune rheumatic disease. J Rheumatol. 2012 Jan;39(1):167-73. doi: 10.3899/jrheum.110721. Epub 2011 Nov 15. PMID 22089462
- [Background] Borba EF, Saad CG, Pasoto SG, Calich AL, Aikawa NE, Ribeiro AC, Moraes JC, Leon EP, Costa LP, Guedes LK, Silva CA, Goncalves CR, Fuller R, Oliveira SA, Ishida MA, Precioso AR, Bonfa E. Influenza A/H1N1 vaccination of patients with SLE: can antimalarial drugs restore diminished response under immunosuppressive therapy? Rheumatology (Oxford). 2012 Jun;51(6):1061-9. doi: 10.1093/rheumatology/ker427. Epub 2012 Jan 31. PMID 22298793
- [Result] Korsun N, Angelova S, Trifonova I, Tzotcheva I, Mileva S, Voleva S, Georgieva I, Perenovska P. Predominance of influenza A(H3N2) viruses during the 2016/2017 season in Bulgaria. J Med Microbiol. 2018 Feb;67(2):228-239. doi: 10.1099/jmm.0.000668. Epub 2018 Jan 3. PMID 29297852
- [Result] Chiu SS, Kwan MYW, Feng S, Wong JSC, Leung CW, Chan ELY, Chan KH, Ng TK, To WK, Cowling BJ, Peiris JSM. Influenza Vaccine Effectiveness Against Influenza A(H3N2) Hospitalizations in Children in Hong Kong in a Prolonged Season, 2016/2017. J Infect Dis. 2018 Apr 11;217(9):1365-1371. doi: 10.1093/infdis/jiy027. PMID 29346614
- [Result] Skowronski DM, Chambers C, De Serres G, Dickinson JA, Winter AL, Hickman R, Chan T, Jassem AN, Drews SJ, Charest H, Gubbay JB, Bastien N, Li Y, Krajden M. Early season co-circulation of influenza A(H3N2) and B(Yamagata): interim estimates of 2017/18 vaccine effectiveness, Canada, January 2018. Euro Surveill. 2018 Feb;23(5):18-00035. doi: 10.2807/1560-7917.ES.2018.23.5.18-00035. PMID 29409570
- [Derived] Aikawa NE, Borba EF, Balbi VA, Sallum AME, Buscatti IM, Campos LMA, Kozu KT, Garcia CC, Capao ASV, de Proenca ACT, Leon EP, da Silva Duarte AJ, Lopes MH, Silva CA, Bonfa E. Safety and immunogenicity of influenza A(H3N2) component vaccine in juvenile systemic lupus erythematosus. Adv Rheumatol. 2023 Nov 28;63(1):55. doi: 10.1186/s42358-023-00339-7. PMID 38017564
- [Derived] Claudino Formiga FF, Silva CA, Pedrosa TDN, Aikawa NE, Pasoto SG, Garcia CC, Capao ASV, Martins VAO, Proenca ACT, Fuller R, Yuki EFN, Vendramini MBG, Rosario DCD, Brandao LMKR, Sartori AMC, Antonangelo L, Bonfa E, Borba EF. Influenza A/Singapore (H3N2) component vaccine in systemic lupus erythematosus: A distinct pattern of immunogenicity. Lupus. 2021 Oct;30(12):1915-1922. doi: 10.1177/09612033211040371. Epub 2021 Aug 28. PMID 34459317